CLINICAL TRIAL: NCT05543512
Title: An Allergen-specific Immune Signature-directed Diet vs Sham Diet for Treatment of Eosinophilic Esophagitis: A Pilot-feasibility Study
Brief Title: The Immune Directed Individualized Elimination Therapy (iDIET) Study
Acronym: iDIET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0500; R01DK132001 (NIH)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis; EoE
Keywords: EoE; Eosinophilic Esophagitis; Diet Therapy
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: Targeted elimination diet therapy versus sham diet elimination therapy
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Individualized Diet Elimination Therapy (Experimental): Subjects in this arm will be assigned an allergen-specific immune signature-directed diet to follow for 8 weeks
  Interventions: Device: Algorithm to diagnose food allergens
- Sham Diet Elimination Therapy (Placebo Comparator): Subjects in this arm will be assigned a sham diet to follow for 8 weeks
  Interventions: Other: Sham diet

INTERVENTIONS:
Device: Algorithm to diagnose food allergens — An algorithm to diagnose food allergens that will drive diet intervention assignment for those in the active arm. Subjects randomized to this group will receive a diet assignment based on results of the algorithm.
  Arms: Individualized Diet Elimination Therapy
Other: Sham diet — Sham diet developed via selecting a random number of foods from a random list of the potential eliminated foods.
  Arms: Sham Diet Elimination Therapy

SUMMARY:
This is a randomized, double blind, sham-controlled, pilot/feasibility trial of individualized dietary elimination treatment.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 fashion to follow an allergen-specific immune signature-directed diet or sham diet during the 8-week treatment period. Blood and biopsies specific to this study will be collected during a baseline endoscopy completed as part of their routine clinical care. Samples will be immediately transported to a lab in which T-cell and immunoglobulin G4 (IgG4) signatures will be analyzed for the full 18 food panel. If randomized to the active intervention, then participants in a blinded fashion will be assigned a diet that removes the foods for which they had a positive threshold result on either the T-cell or IgG4 assay. If randomized to the sham diet, then participants will be provided a sham diet. Sham diets will be developed via selecting a random number of foods from a random list of the potential eliminated foods. The participant, investigators, clinical research coordinators, and study dietician will be blinded to the results of laboratory analysis during the course of the study. The lab, study monitor, or other designee not otherwise involved in the study will be unblinded.

Upon assignment of their diet intervention, participants will meet with a study dietician to discuss their baseline food consumption and assigned diet intervention. After 4 and 8 weeks of diet intervention, they will check-in with the study dietician. In addition, they will monitor their food intake for compliance. At the end of the 8-week treatment period, participants will return for an endoscopy with biopsies and blood draw. Upon completion of the 8-week endoscopy, participation in this study is complete and participants will return to routine care of their condition which may include dietary re-introduction if clinically indicated after completion of the iDIET study.

The primary hypothesis is that participants treated with the immune-signature diet will have significantly lower post-treatment eosinophil counts and dysphagia symptom scores than participants treated with sham diet.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Age: 16 - 80 years
* Diagnosis of EoE as per consensus guidelines
* No prior treatment with, or documented failure of, dietary elimination therapy. Failure is defined as =>15 eos/hpf after a course of the six-food elimination diet (SFED).
* On stable diet for 4 weeks prior to screening endoscopy and agree to maintain throughout course of participation. Foods eliminated for allergic or other reactions are not exclusionary and may continue to be avoided throughout participation in the study regardless of food trigger results.

In addition to meeting the above criteria, to be eligible for randomization an individual must meet all of the following criteria:

* Active EoE (=>15 eos/hpf) based on clinical biopsies taken during baseline endoscopy
* Must have at least one positive food on the IgG4 or T cell stimulation assay

Exclusion Criteria:

* Concomitant eosinophilic gastritis and/or enteritis, confirmed with a prior clinicohistologic diagnosis
* Use of systemic corticosteroids within 4 weeks of the baseline/qualifying endoscopic exam
* Previous esophageal resection
* History of bleeding disorder or esophageal varices
* Current use of blood thinners such as coumadin, warfarin, heparin, and/or novel anticoagulant agents (requires discontinuation of medication within an appropriate time frame for that specific agent and in accordance with standard clinical practice)
* Medical instability that precludes safely performing upper endoscopy
* Inability to read or understand English
* Pregnancy or breastfeeding
* Body mass index (BMI) <17

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Post-treatment peak eosinophil count | 8 weeks
  Post-treatment peak eosinophil count (measured in eos/hpf)

SECONDARY OUTCOMES:
Dysphagia symptom score | 8 weeks
  Dysphagia symptom score, as measured by the validated Eosinophilic Esophagitis Activity Index (EEsAI) instrument This score ranges from 0-100, with higher scores indicating more severe symptoms. A score of < 20 indicates clinical remission.
Endoscopic severity | 8 weeks
  Endoscopic severity will be assessed using the validated EoE Endoscopic Reference Score (EREFS). This score measures endoscopic severity with a set of five endoscopic findings (exudates, rings, edema, furrows, and strictures), and ranges from 0-9, with higher scores indicating higher endoscopic severity.
Percentage of Histologic Responders | 8 weeks
  Histologic response is defined as an esophageal eosinophil count of <15 eos/hpf, a threshold previously determined to be optimal for response assessments in EoE studies

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT05543512/ICF_000.pdf